CLINICAL TRIAL: NCT02500667
Title: A Phase 1, Open-label, Drug-Drug Interaction Study to Assess the Steady State Pharmacokinetics of N91115 Alone and in the Presence of Multiple Dose Administration of Rifampin in Healthy Adult Subjects (SNO-5)
Brief Title: A Drug-Drug Interaction Study of N91115 +/- Rifampin in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nivalis Therapeutics, Inc. (Industry)
Collaborators: Davita Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N91115-1H-04 (SNO-5)
Record Dates: First submitted 2015-07-10; First posted 2015-07-16 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Drug Interaction Potentiation
Keywords: N91115; Rifampin; drug interaction; Cavosonstat
MeSH Terms: interventions — cavosonstat; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- N91115 + Rifampin (Experimental): N91115 200 mg twice daily (BID) from Study Day 1- 13, Rifampin 600 mg once daily (QD) from Study Day 8 - 12
  Interventions: Drug: N91115; Drug: Rifampin

INTERVENTIONS:
Drug: N91115 — 200 mg BID
  Other Names: Cavosonstat
Drug: Rifampin — 600 mg QD
  Other Names: Rifadin

SUMMARY:
The present study is designed to assess the effects of Rifampin on the pharmacokinetics of N91115 in healthy subjects.

DETAILED DESCRIPTION:
This study will assess the effects of multiple oral dose administration of rifampin on the steady state plasma pharmacokinetics (PK) of N91115 in healthy subjects.

Eligible subjects (n=15) will receive oral doses of N91115 twice daily (approximately every 12 hours) on Study Days 1 through the morning of Day 13. On Study Days 8 through 12, rifampin administered 600 mg once daily will be added to the N91115 regimen. Study subjects will be monitored for safety while housed in the clinical research unit (CRU) until discharge on Day 14. Pharmacokinetics will be followed from Study Day 1 through Study Day 14. A follow-up phone call will be made on Day 20 (1 day). Participation of an individual subject may last up to approximately 48 days from the time of screening until the end-of-study follow-up call.

ELIGIBILITY:
Inclusion Criteria:

* Subject voluntarily agrees to participate in this study; signs an IRB-approved informed consent
* Subject is healthy as determined by the screening medical evaluation (including but not limited to medical history, physical examination and clinical laboratory evaluations)
* Subject is Caucasian
* Female subject must be of non-childbearing potential or post-menopausal
* Male subject must agree to use a condom with spermicide and refrain from sperm donation from Day -1 until 30 days post last dose or have a vasectomy at least 6 months prior to screening
* Subject is a non-smoker
* Subject has a body weight > 45 kg and BMI between 18 and 32 kg/m2
* Subject has no clinically significant vital signs finding at screening or Day -1, per the investigator's judgment
* Subject has no clinically significant abnormal findings in 12-lead ECG , per the investigator's judgment, at screening

Exclusion Criteria:

* Subject has clinically significant history or evidence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological, or psychiatric disorder(s)
* Subject has abnormal 12-lead ECG at screening per protocol
* Subject has any disorder that would interfere with the absorption, distribution, metabolism or excretion of drugs
* Subject has any concurrent disease or condition that, in the opinion of the investigator, would make the subject unsuitable for participation in the clinical study
* Subject is a current alcohol abuser and/or has a history of illicit drug abuse within 1 year prior to dosing
* Subject has a positive screening test for Hepatitis B surface antigen, Hepatitis C antibody, or human immunodeficiency virus (HIV) antibody
* Subject is unwilling to refrain from consumption of coffee and caffeine-containing foods and beverages from Day -1 until discharge on Day 14
* Subject is unwilling to abstain from using alcohol beverages from Day -1 until discharge on Day 14
* Subject has donated blood (> 500 mL) or blood products within 56 days prior to Day -1
* Subject has used over-the-counter (OTC) medications (including vitamins) from Day -7, or prescription medications, or herbal remedies from Day -14 until end-of-study follow-up call. By exception, acetaminophen ≤ 1000 mg/day is permitted except within 48 hours prior to Day -1 and hormone replacement therapy (HRT) is allowed throughout the study
* Subject has used an investigational drug within 30 days prior to Day 1 dosing
* Subject has a history of bleeding disorders

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Assess the Potential Effects of Rifampin on N91115 Steady State Area Under the Curve (AUC) Values | On Study Day 14
  To assess the effects of multiple oral dose administration of rifampin on the steady state AUC on Day 14 of N91115 in healthy subjects.

SECONDARY OUTCOMES:
Effects of Rifampin on the AUC vs time of Metabolites of N91115 | On Study Day 14
  make a preliminary non statistical assessment on the effects of multiple oral dose administration of rifampin on steady state plasma PK of N91288 and metabolites, in healthy subjects
The number of participants with adverse events | Over the 21 days of the study
  To evaluate the safety and tolerability of multiple oral doses of N91115 in the presence and absence of multiple oral doses of rifampin
Effects of Rifampin on N91115 and its Metabolites on Urine 12 Hour drug concentrations | Day 14 assessment
  To make a preliminary non statistical assessment on the effects of multiple oral dose administration of rifampin on the 12 hour steady state urine PK of N91115 and its primary metabolites in healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Galloway, MD, Principal Investigator — Davita Clinical Research
Locations (1):
- St. Anthony's Medical Plaza 1, Lakewood, Colorado, United States

REFERENCES:
- [Derived] Donaldson SH, Solomon GM, Zeitlin PL, Flume PA, Casey A, McCoy K, Zemanick ET, Mandagere A, Troha JM, Shoemaker SA, Chmiel JF, Taylor-Cousar JL. Pharmacokinetics and safety of cavosonstat (N91115) in healthy and cystic fibrosis adults homozygous for F508DEL-CFTR. J Cyst Fibros. 2017 May;16(3):371-379. doi: 10.1016/j.jcf.2017.01.009. Epub 2017 Feb 13. PMID 28209466